CLINICAL TRIAL: NCT02824978
Title: Therapeutic Alliance is it Associated With Better Compliance Amongst Children With Juvenile Idiopathic Arthritis ?
Acronym: ALLIANCE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ALLIANCE (RB 16.004 )
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Juvenile Idiopathic Arthritis
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
to evalute if therapeutic alliance is related to adherence in JIA

DETAILED DESCRIPTION:
The therapeutic alliance is the agreement that is being built between doctor and patient during the construction process of care. So active collaboration based on a shared assessment of issues and agreement on possible solutions. Initially described in psychiatry, this analytical concept has been extended to several chronic diseases in particular requiring more often a strong link between doctor and patient. His measure is important since it has been demonstrated by several previous studies that the therapeutic alliance is predictive of the therapeutic effects of treatment. This alliance, however, was little studied in juvenile idiopathic arthritis, its connection with the observance or the quality of life has never been evaluated.

The chronic nature of juvenile idiopathic arthritis (JIA) requires a strong ability of the child to follow his treatment, where the role of parents going to be important and where the relationship built with the caregiver is also essential.

Adherence is a complex concept for which there is no ideal measure. Direct evaluation criteria such as bioassays prove still incomplete and difficult to implement in observational studies. Indirect measures have been developed through self-administered questionnaires and literature showed their relatively good correlation with actual catches. The innovative hypothesis of this research is that a better therapeutic alliance is associated with better adherence child in JIA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with JIA (see classification above)
* Aged at least 8 to 18 years.
* Having already seen more than 2 times in consultation with the referring physician will even include the child in the study so that the alliance could build process
* Children can read, understand and complete questionnaires
* No opposition made

Exclusion Criteria:

* Systemic form of JIA;
* Children aged under 8 years old or over 18 years;
* Child or parent does not understand French
* Refusal of participation

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with Juvenile idiopathic arthritis (JIA) and aged from 8 to 18 years, that have been akready seen more than 2 times in consultation by the same practitioner.
  Treatment is based on the non-steroidal anti-inflammatory drugs, corticosteroids or immunosuppressant therapy and due to chronic nature of JIA, it requires a strong ability of the child to follow his treatment. The role of parents going to be important and the relationship built with the caregiver is essential. As much as in adults, and can be more complex way the question of adherence / therapeutic adherence.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Relationship between therapeutic alliance and compliance judged by the child ( CarQ Questionnaire) and parent ( PARQ Questionnaire). | at inclusion
  Several questionnaires (6-8) measure the alliance in adults and have shown the link between early alliance and therapeutic efficacy and especially the need to measure not made by the therapist but by the treatment. Then the scores were developed in children where the alliance is special since the role of the adult, the parent is part of the monitoring and assistance to the acceptance of the disease and guarantee the continuity of care . Among them, the HQA I was designed to examine the child-parent-caregiver triad. The HQA-CP score (Helping questionnaires Alliance for Child and Parents) is derived from this score. HQA-CP was validated in French by Kermarrec et al.

SECONDARY OUTCOMES:
Quality of Life (CHAQ Questionnaire ) | at inclusion
  The quality of life related to health is important to consider in children in JIA. It can be modified by the treatment, and many other non-medical factors, some limit adherence. Research has shown that better adherence to treatment was associated with a better quality of life. The quality of life is typically measured by the validated CHAQ in French since 2001. It includes 30 items divided into eight areas rated from 0 to 3. It has been validated for different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Devauchelle-Pensec, Professor, Principal Investigator — University Hospital, Brest
Locations (17):
- France (17):
  - CHU Angers, Angers
  - Hôpital Nord Franche Comté, Belfort
  - CHRU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - Hôpital Femme-Mère-Enfant - HCL, Bron
  - CHU Dijon, Dijon
  - CHU Martinique, Fort-de-France
  - Hôpital Bicêtre - APHP, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - CH Mulhouse, Mulhouse
  - CHU Nîmes, Nîmes
  - Hôpital Necker-Enfants Malades - APHP, Paris
  - CHU Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHRU Strasbourg, Strasbourg
  - CHU Nancy, Vandœuvre-lès-Nancy